CLINICAL TRIAL: NCT01579864
Title: Interventional Rigid Bronchoscopy Under General Anesthesia: Influence of the Muscle Relaxant, Succinylcholine or Rocuronium, on the Quality of the Surgical Procedure
Brief Title: Succinylcholine or Rocuronium for Rigid Bronchoscopy Under General Anesthesia
Acronym: Broncho-SR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recent publication (Ghezel-Ahmadi. Thorac Cardiovasc Surg. 2014 Nov 21)
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/05; 2011-000370-59 (EudraCT Number)
Record Dates: First submitted 2012-01-04; First posted 2012-04-18 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Anesthesia
MeSH Terms: interventions — Succinylcholine; Rocuronium

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- succinylcholine (Active Comparator): Succinylcholine 1 mg/kg and a second dose if necessary.
  Interventions: Drug: succinylcholine
- Rocuronium (Experimental): rocuronium 0,9 mg/kg with additional boluses of 0,3 mg/kg f necessary
  Interventions: Drug: rocuronium

INTERVENTIONS:
Drug: succinylcholine — Succinylcholine 1 mg/kg and a second dose if necessary. Rocuronium 0,4 mg/kg can be used as a rescue
  Arms: succinylcholine
Drug: rocuronium — rocuronium 0,9 mg/kg with additional boluses of 0,3 mg/kg f necessary
  Arms: Rocuronium

SUMMARY:
Myorelaxation is generally used as a part of general anesthesia for interventional rigid bronchoscopy. Succinylcholine is most often used because its short duration of action but rocuronium can be used since sugammadex permits a rapid and complete reversal of the neuromuscular block. The aim of ths study is to compare both agents.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for an interventional rigid bronchoscopy under general anesthesia

Exclusion Criteria:

* pregnant woman or woman of childbearing age,
* morbid obesity,
* drug allergy,contra-indication to succinylcholine, rocuronium, sugammadex, propofol, remifentanil,
* history of central neurological or brain damage,
* psychotropic treatment,
* pacemaker,
* renal failure,
* disease of the neuromuscular junction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Score of quality of the surgical procedure | one day
  The quality of the surgical procedure is evaluated by the surgeon (composite score) who is unaware of the neuromuscular agent used (see Fuchs-Buder et al. Acta Anaesthesiol Scand 2007;51(7):789-808)

SECONDARY OUTCOMES:
Score of quality of anesthesia | one day
  The quality of anesthesia is evaluated by the anesthesist in charge on a scale 0-30 (0-10 for the induction ; 0-10 for maintenance; 0-10 for recovery)

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Le Guen, MD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, Île-de-France Region, France